CLINICAL TRIAL: NCT06141967
Title: Evaluating of the Impact of a Connected and Non-intrusive Device in Improving the Screening of Sleep Apnea Syndrome and the Addressing of Potentially Pathological Patients in Hospital Environment
Acronym: AMELIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23CH133; ANSM (Other: 2023-A01288-37)
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea Syndromes; Metabolic Syndrome; Diabetes; Obese
Keywords: Sleep Apnea Syndromes; Diabetes; Withings Sleep analyzer; Epworth; Berlin
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WITHINGS Sleep Analyzer (Experimental): The sleep apnea screening device used is a medical screening device WITHINGS Sleep Analyzer (WSA)
  Interventions: Device: WITHINGS Sleep Analyzer

INTERVENTIONS:
Device: WITHINGS Sleep Analyzer — Potentially eligible patients will be offered to participate in the study, the information leaflet will be given to them and the informed consent form will be signed if the patient agrees to participate in the study.
  In hospitalization in Endocrinology:
  * Realization of the current care report
  * Including systematic achievement of EPWORTH and BERLIN scores
  * Activation of the WSA throughout the duration of the hospitalization
  * Completion of a feasibility questionnaire for the team
  * Quantification of the non-usable screening technique
  * Completion of a patient experience questionnaire at the end of the stay
  * In the event of published positive criteria either for the BERLIN questionnaires, EPWORTH questionnaires or WSA, the patient will be referred to the VISAS center for definitive diagnostic evaluation by polygraphy or polysomnography.
  Other Names: WSA

SUMMARY:
Diabetes, obesity and metabolic syndrome are closely linked to sleep apnea syndrome. Indeed, diabetic and/or obese patients present an increased risk of sleep apnoea syndrome (SAS), with a prevalence estimated at between 10 and 22%, depending on the study, and most of them requiring treatment with Continuous Positive Airway Pressure (CPAP). In this sub-population of patients, only between 40% and 50% benefit from CPAP.

DETAILED DESCRIPTION:
There is therefore an under-referral of diabetic patients to treatment, perhaps linked to the way care is organized, which clogs up the circuit and slows down or even prevents access to care. The investigators would like to test a new organization of care to facilitate and intensify this screening.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years old
* Diabetes Mellitus (Type 1 or 2), or obesity (BMI>30kg/m²) or metabolic syndrome
* Hospitalized for at least one night in the Endocrinology department
* Affiliated or entitled to a social security scheme
* Having received informed information about the study and having co-signed, with the investigator, the informed consent form for participation in the study

Exclusion Criteria:

* Known and/or treated OSAS-type respiratory pathology
* No signature of the informed consent form
* Minor or adult patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
patients real positive for each screening technique | Day 2
  Percentage of patients real positive for each screening technique: BERLIN and EPWORTH score and Withings Sleep Analyzer addressed for polysomnography

SECONDARY OUTCOMES:
Number of tests | Day 2
  Number of positive tests / Number of analyzable test for screening for each type of test
Patient's experience with the use of Withings Sleep Analyzer | Day 2
  Patients' experience is evaluated using a questionnaire with the following possible answers: yes a lot, yes a little, not at all.
Nurse's satisfaction with the use of Withings Sleep Analyzer | 3 months
  Nurse's satisfaction is evaluated using a questionnaire with the following possible answers: yes a lot, yes a little, not at all.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha GERMAIN, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No